CLINICAL TRIAL: NCT03324958
Title: VIrtual REality Glasses for the Enhancement of Acute BRACHYtherapy Tolerance for Endometrial Cancer Patients.
Acronym: Vire-Brachy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment difficulties
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other); Centre Antoine Lacassagne (Other); Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-0501; 2017-A01919-44 (Other: ANSM)
Record Dates: First submitted 2017-10-20; First posted 2017-10-30 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer; Brachytherapy; Virtual reality; Pain; Anxiety
MeSH Terms: conditions — Endometrial Neoplasms; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Assessment of the mean local pain during brachytherapy applicator'setting up, with and without virtual reality helmet use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Helmet (Experimental): Patients will use a virtual reality helmet during brachytherapy applicator's setting up. The use of virtual reality helmet has already been assessed during oncologic treatments, and seems to reduce pain and anxiety. The use of virtual reality helmet has never been assessed to reduce the pain or anxiety associated with brachytherapy applicators' setting up.
  Interventions: Device: Virtual reality Helmet
- No Virtual Reality Helmet (Active Comparator): Patient wont use virtual reality helmet during brachytherapy applicator setting up, as in current practice.
  Interventions: Other: No Virtual Reality Helmet

INTERVENTIONS:
Device: Virtual reality Helmet — The virtual reality helmet will be installed by a radiotherapist or a radiotherapy manipulator, just before the intra vaginal applicator. The virtual reality headset will be connected to a dedicated computer. The virtual reality program will run for 10 minutes which will cover the entire procedure for setting up the brachytherapy device. In order to optimize the distractive potential of virtual reality, four different virtual reality programs will be offered to patients during each brachytherapy fraction. These programs will be contemplative so as not to compromise the immobility of the patients during the installation of the brachytherapy applicator.
  Arms: Virtual Reality Helmet
Other: No Virtual Reality Helmet — The radiotherapists can freely dialogue with the patients during the brachytherapy applicator' seating up, as in current practice.
  Arms: No Virtual Reality Helmet

SUMMARY:
This randomized phase III multicenter trial aims to evaluate the impact of virtual reality helmets (visual and audio) during VCB in patients treated for endometrial cancer, in terms of pain and anxiety.

DETAILED DESCRIPTION:
Endometrial cancer is one of the most common gynaecological cancers among women in the developed countries. After a curative surgical treatment, many relapses occur in the vaginal cuff. The PORTEC-2 trial has demonstrated a similar reduction in local relapses of intermediate- to high-risk endometrial cancer with vaginal cuff brachytherapy (VCB) than with external beam radiotherapy (EBRT). However, VCB induced less late toxicities. VCB is therefore indicated after surgery for intermediate- to high-risk endometrial cancer. VCB is also recommended after radiation therapy, for patients with stage II or III type 1 endometrial cancers according to the International Federation of Gynaecology and Obstetrics classification (FIGO), and for all patients with histological type 2 endometrial cancers.

If the late tolerance of VCB is correct, the acute tolerance remains limited, and is mainly characterized by local pain and anxiety) Virtual reality appears to be a promising tool to enhance treatment cancer tolerance, offering a safe and entertaining environment. By the way, the use of virtual reality could limit physical and psychical discomfort induced by VCB.

This randomized phase III multicenter trial aims to assess the impact of virtual reality helmets (visual and audio) during VCB in patients treated for endometrial cancer, in terms of pain (primary endpoint), and in terms of anxiety (secondary endpoint). Randomization will define which patient will wear a virtual reality helmet. Stratification will be performed according to the following criteria: vaginal molded applicator versus cylinder, two applications versus four; <70 years versus> 70 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* Patients with endometrial cancer, with histological type I and II, regardless of the degree of differentiation.
* Patients with stage I, II or III endometrial cancer according to the FIGO classification.
* Patients treated with high-dose-rate vaginal cuff brachytherapy, with curative intent.
* Patients affiliated or entitled to a social security scheme.
* Patients who received information about the study and co-signed with the investigator the consent to participate at the study.

Exclusion Criteria:

* Patients with stage IV endometrial cancer according to FIGO classification.
* Patients presenting recurrence of endometrial cancer.
* Pregnant or nursing women.
* Patients under protection of justice or unable to give consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Mean pain during brachytherapy applicator installations | 1 week
  Pain assessment will be done with visual analogue scale pain (line of 10 centimeters without graduation : beginning of the line means no pain, and the terminal extremity means worst pain ever felt), before and after brachytherapy applicator setting up

SECONDARY OUTCOMES:
Pain during brachytherapy applicator installations, independently at each fraction | 1 week
  Pain assessment will be done with visual analogue scale pain (line of 10 centimeters without graduation : beginning of the line means no pain, and the terminal extremity means worst pain ever felt), before and after brachytherapy applicator setting up.
Mean anxiety during brachytherapy applicator installations | 1 week
  Anxiety assessment will be done with visual analogue scale (line of 10 centimeters without graduation : beginning of the line means no pain, and the terminal extremity means worst pain ever felt) anxiety, before and after brachytherapy applicator setting up, and with Hamilton scale (scores will be comprised between 0 : no anxiety, and 30 : maximal anxiety) before brachytherapy applicator setting up.
Quality of life, six to height weeks after brachytherapy | 6 to 8 weeks after brachytherapy
  Quality of life assessment will be done with the the endometrial cancer (EC)-specific Quality of Life module of the European Organization for Research and Treatment of Cancer (EORTC QLQ-EN24).
Anxiety and depression, six to height weeks after brachytherapy | 6 to 8 weeks after brachytherapy
  Anxiety and depression will be assessed six to height weeks after brachytherapy with the Hamilton Anxiety and Depression scale (scores will be comprised between 0 : no anxiety, and 30 : maximal anxiety).
Correlation between mean pain during brachytherapy applicator setting up and age | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and age.
Correlation between mean pain during brachytherapy applicator setting up and G8 scale. | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and G8 scale.
Correlation between mean pain during brachytherapy applicator setting up and histologic type of cancer. | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and histologic type of cancer.
Correlation between mean pain during brachytherapy applicator setting up and FIGO stage. | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and FIGO stage.
Correlation between mean pain during brachytherapy applicator setting up and Performance status. | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and Performance status.
Correlation between mean pain during brachytherapy applicator setting up and patient weight. | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and patient weight.
Correlation between mean pain during brachytherapy applicator setting up and marital status. | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and marital status.
Correlation between mean pain during brachytherapy applicator setting up and socio educational status | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and socio educational status.
Correlation between mean pain during brachytherapy applicator setting up and number of pregnancies. | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and number of pregnancies.
Correlation between mean pain during brachytherapy applicator setting up and history of pelvic surgery | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and history of pelvic surgery.
Correlation between mean pain during brachytherapy applicator setting up and the number of concomitant treatment. | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and the number of concomitant treatment.
Correlation between mean pain during brachytherapy applicator setting up and the nature of concomitant treatment. | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and the nature of concomitant treatment.
Correlation between mean pain during brachytherapy applicator setting up and the nature of cancer treatments | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and the nature of cancer treatments.
Correlation between mean pain during brachytherapy applicator setting up and the supportive cares performed | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and the supportive cares performed.
Correlation between mean pain during brachytherapy applicator setting up and the radiotherapy scheme | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and the radiotherapy achievement
Correlation between mean pain during brachytherapy applicator setting up and the brachytherapy scheme | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and the brachytherapy scheme
Correlation between mean pain during brachytherapy applicator setting up and the radiotherapy induced toxicities (describe according to the Common Terminology Criteria for Adverse Events 4.4) | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and the radiotherapy induced toxicities (describe according to the Common Terminology Criteria for Adverse Events 4.4).
Correlation between mean pain during brachytherapy applicator setting up and the toxicities of previous brachytherapy fractions (describe according to the Common Terminology Criteria for Adverse Events 4.4). | 1 week
  Correlation will potentially be established between pain during brachytherapy applicator setting up and the brachytherapy induced toxicities (describe according to the Common Terminology Criteria for Adverse Events 4.4).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Magné, PhD, Principal Investigator — Institut de Cancérologie Lucien Neuwirth
Locations (2):
- France (2):
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No